CLINICAL TRIAL: NCT06837727
Title: Left Ventricular Outflow Tract Mean Velocity in Children: a Strong Alternative to Cardiac Index in Pediatric Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GIROUX Nathan, Hospital Practitioner, Senior Physician, Central Hospital, Nancy, France
Other Study IDs: 2025PI012
Record Dates: First submitted 2025-02-11; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Shock Circulatory; Cardiogenic Shock
Keywords: Cardiac Index; hemodynamic; echocardiography; intensive care unit
MeSH Terms: conditions — Shock; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Objectives: Noninvasive assessment of cardiac index (CI) in pediatric critical ill patient is crucial. Aortic Velocity Time Integral (VTI) valuable in adults, faces age and heart rate variability challenges in pediatrics, complicating CI interpretation in shocked patients. Measurement errors can complicate CI evaluation, particularly in shocked patients. Considering the proportional relationship between aortic annulus and Body Surface Area (BSA) in children, along with the relatively constant mean aortic velocity, we studied if Left Ventricular Outflow Tract mean-velocity (LVOTmv) reliably estimates bedside CI.

Design : retrospective, observational, single-center study.

Setting : Pediatric Intensive Care Unit (PICU) in a tertiary care hospital.

Patients : one hundred forty-four children in PICU (age 0-17 years, BSA 0.11-1.69 m2) requiring hemodynamic evaluation.

Intervention : Bedside ultrasound by expert cardiologists

Measurements and Main Results : We explored the correlation between LVOTmv (measured in pulse wave doppler from the apical five-chamber view) and standard CI estimation (multiplying aortic VTI, heart rate, and aortic valve area). We excluded arrhythmia and anomalies of the left ventricular outflow tract.

ELIGIBILITY:
Inclusion Criteria:

* infants, children, and adolescents hospitalized in our Pediatric Intensive Care Unit (PICU) in a non-surgical cardiology unit requiring hemodynamic assessment

Exclusion Criteria:

* documented irregular heart rates (HR) or with congenital heart malformations that could affect aortic measurements or LVOT velocity (such as aortic valve anomalies)

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: infants, children, and adolescents hospitalized in our Pediatric Intensive Care Unit (PICU) in a non-surgical cardiology unit
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
correlation between LVOT mean velocity (LVOTmv) from the traditional apical five-chamber view and standard CI measurements | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU of Nancy, Vandœuvre-lès-Nancy, Lorraine, France